CLINICAL TRIAL: NCT01901276
Title: The Effects of Gastric Acid Suppression on the Colonic Microbiome
Brief Title: Effects of Gastric Acid on Colonic Microbiome
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Daniel Freedberg, MD (Other)
Responsible Party: Sponsor-Investigator, Daniel Freedberg, MD, Assistant Professor of Medicine, Columbia University
Organization: Columbia University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: AAAL3307
Record Dates: First submitted 2013-07-12; First posted 2013-07-17 (Estimated); Results first posted 2024-08-15 (Actual); Last update posted 2024-08-15 (Actual); Status verified 2024-07

CONDITIONS: Clostridium Difficile
Keywords: Proton Pump Inhibitors; Microbiome; Clostridium difficile
MeSH Terms: interventions — Omeprazole; BID protein, human

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Omeprazole 40 mg bid x 4-8 weeks (Experimental): See study description for further details.
  Interventions: Drug: Omeprazole 40 mg bid

INTERVENTIONS:
Drug: Omeprazole 40 mg bid — As above.
  Other Names: Brand name: Prilosec

SUMMARY:
The colonic microbiome is essential in human health and disease. Clostridium difficile-associated diarrhea (CDAD), a highly morbid form of infectious diarrhea, is caused by antibiotics which perturb the microbiome and allow C. difficile to proliferate. Proton pump inhibitors (PPIs) are powerful suppressors of gastric acid and among the most common medicines in the United States. Dozens of observational studies show that longterm PPI use is associated with CDAD. However, the mechanism by which PPIs cause CDAD is unknown. We believe that PPIs cause CDAD by inducing alterations in the human colonic microbiome. We will confirm or refute the hypothesized mechanism for the association between PPIs and CDAD using an unblinded, single-armed study design. We will use pyrosequencing of the hypervariable V4 region of the bacterial 16S ribosomal subunit gene in human fecal samples to describe the colonic flora. We will collect fecal samples from volunteers before and after PPIs given for different durations and test the microbiome to determine 1) whether PPIs diminish overall diversity, 2) whether PPIs diminish relative abundance of Bacteroidetes, 3) whether increased duration of PPIs affects diversity, and 4) whether there is recovery of diversity after completing a defined course of PPIs. We believe that PPIs will cause a pattern of diminished overall microbiome diversity and reduced anaerobes - the same pattern seen after use of antibiotics. Furthermore, we believe that increased PPI duration will further diminish diversity and that the microbiome will return to pre-PPI levels of diversity after PPIs are stopped. These results will facilitate biologically-based clinical interventions to reduce rates of CDAD among patients who require acid suppression.

DETAILED DESCRIPTION:
Study Design We will recruit 12 adult volunteers for a crossover study with a total duration of 12 weeks. Subjects will be observed off of PPIs for 4 weeks and then will be placed on PPIs for 4 weeks. Subsequently, subjects will be randomized to receive an additional 4 weeks of PPIs or no therapy. Stool samples will be collected at 4 separate time points.

Study Outcomes and Statistical Analyses The primary outcome will be change in overall diversity of fecal flora after 4 weeks of PPIs compared to 4 weeks of no acid suppression. Additional outcomes to be assessed include the effect of PPIs on the relative abundance of Bacteroidetes at week 4 and change in the diversity of fecal flora at week 8.

ELIGIBILITY:
Inclusion Criteria:

* 18 or more years old
* Able to give informed consent

Exclusion Criteria:

* Use of systemic antibiotics within the past year
* Use of acid suppression medications (PPIs or H2-receptor antagonists) within the past year (antacids permitted if more than one month from date of enrollment)
* History of chronic gastrointestinal mucosal disease (e.g. inflammatory bowel disease, celiac disease, microscopic colitis)
* Any clinically significant or uncontrolled major morbidity, including but not limited to serious cardiac or respiratory disease or uncontrolled HIV
* Abnormal bowel frequency (minimum once every 2 days, maximum 3 times per day)
* Use of clopidogrel or medications with potential significant interaction with PPIs
* Osteoperosis or history of non-traumatic bone fracture
* History of adverse reactions to PPIs
* Initiation of any new medication within the month prior to enrollment
* Pregnancy
* Inability to give informed consent

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2013-08; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Julian A Abrams, MD, MS, Principal Investigator — Columbia University
Locations (1):
- Columbia University, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
Refer to the published study results for summary data.

REFERENCES:
- [Background] Freedberg DE, Toussaint NC, Chen SP, Ratner AJ, Whittier S, Wang TC, Wang HH, Abrams JA. Proton Pump Inhibitors Alter Specific Taxa in the Human Gastrointestinal Microbiome: A Crossover Trial. Gastroenterology. 2015 Oct;149(4):883-5.e9. doi: 10.1053/j.gastro.2015.06.043. Epub 2015 Jul 9. PMID 26164495

RESULTS

PARTICIPANT FLOW:
Groups:
- Omeprazole 40 mg Bid: Participants will take Omeprazole 40 mg twice daily for 4 weeks.
- No Treatment: Participants will not receive a study intervention.
Period: No PPI: Week 0 to Week 4
Arm/Group | Omeprazole 40 mg Bid | No Treatment
Started | 0 | 14
Completed | 0 | 12
Not Completed | 0 | 2
Not completed — Withdrawal by Subject | 0 | 2
Period: On PPI: Week 4 to Week 8
Arm/Group | Omeprazole 40 mg Bid | No Treatment
Started | 12 | 0
Completed | 12 | 0
Not Completed | 0 | 0
Period: Randomization: Week 8 to Week 12
Arm/Group | Omeprazole 40 mg Bid | No Treatment
Started | 6 | 6
Completed | 6 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Healthy volunteers.
Arm/Group | Omeprazole 40 mg Bid x 4-8 Weeks
Number analyzed (Participants) | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 40 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 9
Region of Enrollment [Number; unit: participants]
  United States | 12

OUTCOME MEASURES:

1. Primary Outcome: Shannon Diversity Index Measuring Change in Microbiome Diversity
Description: In order to assess the diversity of the colonic microbiome, the Shannon diversity index will be calculated for each subject:
  * After four weeks of no acid suppression (Week 0 vs. Week 4)
  * After four weeks of twice daily PPI (Week 4 vs. Week 8)
  The Shannon diversity index is a mathematical measure of species diversity in a given community. The Shannon index is calculated as: -∑[(pi)×ln(pi)] where H is the Shannon diversity index, and pi is the proportion of individuals of i-th species in a whole community. The minimum value of the Shannon diversity index is 0, which indicates there's no diversity - only one species is found in that habitat. There is no upper limit to the Shannon index. The higher the value of H, the higher the diversity of species in a particular community.
Time Frame: Baseline (Week 0), Week 4, Week 8
Measure: Median (95% Confidence Interval); unit: Shannon index
Groups:
- Omeprazole 40 mg Bid x 4-8 Weeks: Includes all participants who completed the study.
Arm/Group | Omeprazole 40 mg Bid x 4-8 Weeks
Number analyzed (Participants) | 12
Shannon index
  Change in Shannon indices from Baseline to Week 4 (no PPIs) | 0.18 [-0.32 to 0.68]
  Change in Shannon indices from Week 4 to Week 8 (on PPIs) | 0.14 [-0.23 to 0.51]
Statistical Analysis 1: Comparison: Omeprazole 40 mg Bid x 4-8 Weeks; Within-individual differences in Shannon indices were tested using paired t tests (normally distributed data); Test type: Superiority or Other; p = 0.71, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: Up to 6 months post-intervention.
Groups:
- Omeprazole 40 mg Bid x 4-8 Weeks: See study description for further details. Omeprazole 40 mg bid: As above.
Arm/Group | Omeprazole 40 mg Bid x 4-8 Weeks
All-Cause Mortality (participants affected / at risk) | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No